CLINICAL TRIAL: NCT02646514
Title: Efficacy and Safety of Endobiliary Radiofrequency Ablation by Using a Novel RF Catheter (ELRA®) on Maintaining the Patency of Endobiliary Metal Drainage in Patients With Malignant Biliary Strictures : A Double-arm Comparable Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2015-0053
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Cholangiocarcinoma, Gallbladder Cancer, Pancreatic Cancer
Keywords: Cholangiocarcinoma, radiofrequency ablation, metal stent
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms; Pancreatic Neoplasms | interventions — Radiofrequency Ablation; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RFA with RF catheter (ELRA®) with stenting (Experimental)
  Interventions: Device: Radiofrequency ablation with stenting
- stenting (Active Comparator)
  Interventions: Device: stenting

INTERVENTIONS:
Device: Radiofrequency ablation with stenting — Side viewing endoscope or PTCS scope can be used for all procedures. Cholangiogram is performed to confirm the stricture location, length and diameter. And then, RF catheter (ELRA®) is advanced over a guide wire at the level of the biliary stricture and ablation at 7-10 watts for a time period of 60-120s according to the length is conducted.
  After performance of RFA, metal stents are inserted to ensure adequate decompression and bile drainage.
  Arms: RFA with RF catheter (ELRA®) with stenting
Device: stenting — Metal stents are inserted to ensure adequate decompression and bile drainage. The diameter and stent lengths can be changed according to the lesion.
  Arms: stenting

SUMMARY:
Malignant obstructive jaundice is a common complication of advanced stage cholangiocarcinoma, gallbladder cancer, and pancreatic cancer. In biliary stricture by malignancy, biliary drainage with placement of self-expanding metal stent (SEMS) for palliation is the therapy of choice in these patients. When compared to plastic stents, SEMS present a significantly decreased risk of recurrent biliary obstruction. SEMS are also more cost-effective than plastic stents in patients with a life expectancy of longer than 4 months. However, despite their numerous benefits, SEMS become occluded in up to 50 % of patients in the first 6-8 months.

Radiofrequency ablation (RFA) has been used to treat malignancies of the liver since the early 1990s. Other studies have investigated its role in diseases of the colon and esophagus. More recently, this technique has been recognized for its potential in palliative treatment of malignant biliary strictures. RFA uses a high-frequency alternating current to generate heat and achieve coagulative necrosis when in contact with tissue. Within the bile duct, RFA appears to be safe and may result in decreased benign epithelial hyperplasia and tumor ingrowth. However, RFA along with placement of SEMS has not been well studied. On the other hand, newly developed RFA catheter (ELRA®) showed the feasibility and safety in south korea, recently.

The purpose of this study was to investigate the Efficacy and safety of endobiliary RFA by using a novel RF catheter (ELRA®) on maintaining the patency of endobiliary metal drainage in patients with malignant biliary strictures.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed malignant biliary obstruction or clinically defined malignant biliary obstruction
* older than 19 years old
* Life expectancy > 3 months
* Inoperable case due to advanced stage or comorbidity
* Informed consent

Exclusion Criteria:

* Inadequate case for ERCP
* Inadequate coagulation (platelet count < 60,000/µl, PT(INR)>1.5)
* Abnormal biliary tract system due to previous operation
* Failed endoscopic approach to duodenum or biliary tract
* Pregnancy
* No signed informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Patency of metal stent | 12 months
  Patency of metal stent (From stent insertion date to stent occlusion date or last follow up date if stent is patent)

SECONDARY OUTCOMES:
Overall Survival | 12 months
Complication rate | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sharaiha RZ, Natov N, Glockenberg KS, Widmer J, Gaidhane M, Kahaleh M. Comparison of metal stenting with radiofrequency ablation versus stenting alone for treating malignant biliary strictures: is there an added benefit? Dig Dis Sci. 2014 Dec;59(12):3099-102. doi: 10.1007/s10620-014-3264-6. Epub 2014 Jul 18. PMID 25033929
- [Background] Ortner ME, Caca K, Berr F, Liebetruth J, Mansmann U, Huster D, Voderholzer W, Schachschal G, Mossner J, Lochs H. Successful photodynamic therapy for nonresectable cholangiocarcinoma: a randomized prospective study. Gastroenterology. 2003 Nov;125(5):1355-63. doi: 10.1016/j.gastro.2003.07.015. PMID 14598251
- [Derived] Kang H, Chung MJ, Cho IR, Jo JH, Lee HS, Park JY, Park SW, Song SY, Bang S. Efficacy and safety of palliative endobiliary radiofrequency ablation using a novel temperature-controlled catheter for malignant biliary stricture: a single-center prospective randomized phase II TRIAL. Surg Endosc. 2021 Jan;35(1):63-73. doi: 10.1007/s00464-020-07689-z. Epub 2020 Jun 2. PMID 32488654